CLINICAL TRIAL: NCT00977873
Title: Randomised, Multi-Centre, Double-Blind, Placebo-Controlled Trial of Vitamin D Supplementation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Trial of Vitamin D Supplementation in Chronic Obstructive Pulmonary Disease
Acronym: ViDiCO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-010084-16
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vigantol oil (Active Comparator): Vigantol oil will be administered in 2-monthly oral bolus doses over a period of one year
  Interventions: Dietary Supplement: Cholecalciferol
- Miglyol oil (Placebo Comparator): Miglyol oil will be administered in 2-monthly oral bolus doses over a period of one year
  Interventions: Dietary Supplement: Miglyol oil

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Cholecalciferol will be administered as 2-monthly oral bolus doses of Vigantol oil over a period of one year
  Arms: Vigantol oil
Dietary Supplement: Miglyol oil — Miglyol oil will be administered in 2-monthly bolus doses over a period of one year
  Arms: Miglyol oil

SUMMARY:
The study null hypothesis is that vitamin D supplementation will not influence time to upper respiratory tract infection or time to moderate/severe exacerbation of chronic obstructive pulmonary disease.

ELIGIBILITY:
Principal Inclusion Criteria:

* Medical record diagnosis of COPD, emphysema or bronchitis
* Post-bronchodilator FEV1 / FVC < 70% or post-bronchodilator FEV1 / slow VC < 70%
* Post-bronchodilator FEV1 < 80% predicted
* Age ≥ 40 years on day of first dose of IMP
* Smoking history ≥ 15 pack-years
* If a woman of child-bearing potential, is sexually abstinent or has negative pregnancy test within 7 days of recruitment and agrees to use reliable form of contraception until she has completed the study
* Able to give written informed consent to participate

Exclusion Criteria:

* Current diagnosis of asthma
* Known clinically significant bronchiectasis
* Known sarcoidosis, hyperparathyroidism, nephrolithiasis, active tuberculosis, vitamin D intolerance, liver failure, renal failure, terminal illness, lymphoma or other malignancy not in remission for ≥ 3 years
* Taking benzothiadiazine derivative, cardiac glycoside, carbamazepine, phenobarbital, phenytoin or primidone
* Taking dietary supplement or topical preparation containing vitamin D up to 2 months before first dose of IMP
* Treatment with any investigational medical product or device up to 4 months before first dose of IMP
* Breastfeeding, pregnant or planning a pregnancy
* Baseline corrected serum calcium > 2.65 mmol/L
* Baseline serum creatinine > 125 micromol/L

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to first upper respiratory tract infection | One year
Time to first moderate / severe COPD exacerbation | One year

SECONDARY OUTCOMES:
Time to unscheduled health service use for upper respiratory tract infection or moderate / severe exacerbation of chronic obstructive pulmonary disease | One year
Proportion of participants experiencing hypercalcaemia | One year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian R Martineau, MRCP, Study Director — Queen Mary University of London
Locations (4):
- United Kingdom (4):
  - Lower Clapton Health Centre, London
  - Homerton University Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Barts and The London NHS Trust, London

REFERENCES:
- [Derived] Martineau AR, James WY, Hooper RL, Barnes NC, Jolliffe DA, Greiller CL, Islam K, McLaughlin D, Bhowmik A, Timms PM, Rajakulasingam RK, Rowe M, Venton TR, Choudhury AB, Simcock DE, Wilks M, Degun A, Sadique Z, Monteiro WR, Corrigan CJ, Hawrylowicz CM, Griffiths CJ. Vitamin D3 supplementation in patients with chronic obstructive pulmonary disease (ViDiCO): a multicentre, double-blind, randomised controlled trial. Lancet Respir Med. 2015 Feb;3(2):120-130. doi: 10.1016/S2213-2600(14)70255-3. Epub 2014 Dec 2. PMID 25476069